CLINICAL TRIAL: NCT06814665
Title: EPI-NY: Improving Diagnostics and Care After First Seizure
Brief Title: Improving Diagnostics and Care After First Seizure
Acronym: EPI-NY
Status: Recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 807588
Record Dates: First submitted 2025-01-24; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: First Suspected Epileptic Seizure
Keywords: epilepsy; first seizure; early epilepsy; EEG; AI
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- First epileptic seizure: The patient has experienced one or more first-in-life events with a substantial suspicion of being an epileptic seizure, excluding febrile seizures, and these episodes have previously not been evaluated by a neurologist or pediatrician
- New evaluation of possible seizures previously thought to be non-epileptic: The patient has experienced the recurrence of events with a substantial suspicion of being an epileptic seizure, that have previously been evaluated by a neurologist or pediatrician to not be epileptic, and this merits a new evaluation.
- New epilepsy diagnosis in the study period not otherwise included: The patient does not fulfill the criteria for the two other groups, but has been investigated for episodes or complaints, which after evaluation have been shown to be first-in-life epileptic seizures

SUMMARY:
A first epileptic seizure is a distressing experience, often leading to a complicated and discouraging journey before an epilepsy diagnosis is confirmed. Early diagnostics can help alleviate this uncertainty. It is important to note that seizure mimics and suspected epilepsy are more frequently encountered than an actual first diagnosis of epilepsy or an epileptic seizure. Conversely, delays in diagnosing epilepsy are also common. The current evidence base on first events that may be epileptic remains limited.

First seizure clinics, which provide specialized care for these cases, are becoming more common globally, but none have yet been established in Norway. There is a pressing need to assess the prevalence of first-seizure-like events in Bergen and the surrounding areas, as well as to investigate the clinical trajectory before and after an epilepsy diagnosis. EEG is the cornerstone of diagnostic testing for epilepsy after first seizure, and recent advancements have introduced artificial intelligence to enhance the accuracy of EEG-based epilepsy identification.

The investigators will identify in one year around 200 hospital-handled patients who had had an episode that may be epileptic. Patient will be followed up over two years, with data abstracted from the medical record regarding seizure diagnosis, new events, new brain-related diagnoses and complications. Data will also be gathered from government databases in primary and secondary care regarding complications from seizure, new brain-related diagnoses, new brain-related medications, sickness absence and income. For children, school absence days will be collected.

The investigators will identify the incidence of first seizure and new-onset epilepsy, and and which care pathways most patients with suspected first seizure go through. The investigators will study the role of early EEG to reduce diagnostic uncertainty, and compare conventional EEG interpretation with AI-assisted interpretation for diagnostic precision. The investigators will study the trajectory of anxiety, quality of life and complications with record linkage for epilepsy-relevant outcomes. A broad scope of complications will be studied, including job or school absence, driving license status, injuries in primary or secondary care, and new brain-related diagnoses. This study will gather important data to gauge potential gaps and improvements in care in early epilepsy, of relevance to patients in Bergen, Norway and the developed part of the world.

Particulary novel aspects are an evaluation of the SCORE AI model for EEG analysis, and linking to a spectrum of government databases on work participation, primary care and specialty care on complications of first seizure and/or early epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* The patient has experienced events with a substantial suspicion of being an epileptic seizure. One of:

  * The patient has experienced one or more first-in-life events with a substantial suspicion of being an epileptic seizure, including febrile seizures, and these episodes have previously not been evaluated by a neurologist or pediatrician OR
  * The patient has experienced the recurrence of events with a substantial suspicion of being an epileptic seizure, that have previously been evaluated by a neurologist or pediatrician to not be epileptic, and this merits a new evaluation.
  * OR: The patient does not fulfill the criteria above, but has been investigated for episodes or complaints, which after evaluation have been shown to be first-in-life epileptic seizures.

OR

-The patient has experienced the recurrence of events with a substantial suspicion of being an epileptic seizure, that have previously been evaluated by a neurologist or pediatrician to not be epileptic, and this merits a new evaluation.

Exclusion Criteria:

* Previous known clinical diagnosis of epilepsy given by a neurologist or pediatrician, and not subsequently retracted.
* Person or caregivers able to give informed consent.
* Adequate Norwegian language skills to be able to fill out questionnaires.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: First epileptic seizure, or multiple previous seizures not evaluated by a neurologist or child neurologist
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2027-01-24 (Estimated); Study Completion 2029-01-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of first seizure and new-onset epilepsy | 2 years
  Based on the final two year status, or last-status carried forward, the incidence of first seizures and new-onset epilepsy will be calculated for adults and children.
Percent diagnostic EEG | 2 years
  The diagnostic yield of early vs late yield will be categorized as routine-EEG within 24 hours, or LTM-EEG within 1 week or later. The diagnostic yield will be computed as the percentage of patients with interictal epileptiform discharges or seizure during EEG for each category and time frame for EEG, and the same for final epilepsy diagnosis
Sensitivity, specificity, accuracy of human vs human-AI-assisted EEG analysis to predict future epilepsy | 2 years
  We will compare the results of the current clinical standard of care, which is human expert EEG interpretation, with expert-assisted AI analysis using the SCORE AI model EEG software . We will compute sensitivity, specificity, accuracy for both diagnostic pipelines applied to all EEG to predict a future epilepsy diagnosis taken from medical records, as well as subtype of epilepsy (focal, idiopathic, unknown).
Seizure control in new-onset epilepsy | 2 years
  Among patients with new-onset epilepsy, the percentage suffering no new epileptic seizures will be measured.
Seizure-related trauma | 2 years
  Among patients with new-onset epilepsy, what percentage suffer from seizure-related trauma in the first and subsequent eventscompared to patients with first epileptic seizure without new-onset epilepsy and compared to patients with other event diagnosis in the same time period
Loss of driving license | 2 years
  Among patients with new-onset epilepsy, what percentage suffer from loss of driving license compared to patients with first epileptic seizure without new-onset epilepsy and compared to patients with other event diagnosis in the same time period
Loss of labor market participation | 2 years
  Among patients with new-onset epilepsy, what percentage suffer from loss of labor market participation compared to patients with first epileptic seizure without new-onset epilepsy and compared to patients with other event diagnosis in the same time period
New-onset psychiatric diagnoses | 2 years
  Among patients with first seizure, and new-onset epilepsy, what percentage suffer from new-onset psychiatric diagnoses compared to patients with first epileptic seizure without new-onset epilepsy and compared to patients with other event diagnosis in the same time period

SECONDARY OUTCOMES:
Time to review EEG | 2 years
  The time to review EEG will also be compared between expert vs expert-AI-assisted EEG analysis
QOLIE31 | 2 years
  Adults will be followed longitudinally with self-reported measures of quality of life (QOLIE31)
GAD7 | 2 years
  Adults will be followed longitudinally with self-reported anxiety (GAD7)
Brief COPE | 2 years
  Adults will be followed longitudinally with self-reported coping (Brief COPE)
Kindl | 2 years
  Children will be followed longitudinally with parent-reported quality of life (Kindl)
Mortality | 2 years
  Among patients with first seizure, and new-onset epilepsy, what percentage suffer from mortality compared to patients with first epileptic seizure without new-onset epilepsy and compared to patients with other event diagnosis in the same time period
School absence days | 2 years
  Among children with new-onset epilepsy, what percentage suffer from increased school absence days compared to children with first epileptic seizure without new-onset epilepsy and compared to children with other event diagnosis in the same time period

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brogger, MD PhD, Principal Investigator — Helse-Bergen HF
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
GDPR makes this very difficult